CLINICAL TRIAL: NCT02608567
Title: Prognostic Impact of Myocardial Longitudinal Strain in Asymptomatic Aortic Stenosis: a Meta-Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Association of Cardiovascular Imaging (Other)
Responsible Party: Principal Investigator, Julien Magne, EACVI board member - Research&Innovation committee member, European Association of Cardiovascular Imaging
Other Study IDs: EACVI-001
Record Dates: First submitted 2015-11-17; First posted 2015-11-18 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Aortic Valve Stenosis; Asymptomatic Conditions; Left Ventricular Function
MeSH Terms: conditions — Aortic Valve Stenosis; Asymptomatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preserved LV GLS: Patients will be compared according to the level of LV global longitudinal strain (GLS) as derived from transthoracic echocardiography and speckle tracking analysis.
  Two groups will be compared regarding outcome: preserved LV GLS vs. reduced LV GLS. The definition use for reduced LV GLS will be >-16%. An optimal threshold would also be calculated and derived from the pooled data.
- Reduced LV GLS: The definition use for reduced LV GLS will be >-16%. An optimal threshold would also be calculated and derived from the pooled data.

SUMMARY:
In patients with asymptomatic aortic stenosis (AS), the prognostic value of reduced left ventricular (LV) ejection fraction is well known. Consequently, there is class I indication for surgery in these patients when LV ejection fraction <50%. However, there is growing evidences suggesting that subclinical LV dysfunction, and more particularly longitudinal myocardial dysfunction, may be a powerful early predictor of outcome, even when LV ejection is still preserved. In asymptomatic AS patients with LV ejection fraction >50%, a reduced LV global longitudinal strain, as assessed using speckle tracking imaging with transthoracic echocardiography, may be an accurate marker to identify early subclinical LV dysfunction and thus, to improve the risk stratification, the management and the timing of surgery. Several mono-centric observational small studies recently reported results emphasizing the role of LV global longitudinal strain in AS patients. Therefore, a meta-analysis may be conducted and may provide meaningful data. The investigators hypothesized that LV global longitudinal strain is a determinant of outcome in asymptomatic patients with AS and preserved LV ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* studies selected in PubMed, Embase, Ovid, and Google Scholar, published between 2005 and 2015 without language restriction according to the following criteria: "aortic stenosis" AND "longitudinal strain"

Exclusion Criteria:

* Studies reporting global longitudinal strain derived from VVI and not speckle tracking analysis.
* Studies with cohort of patients with aortic valve replacement indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic patients with at least moderate aortic stenosis (mean pressure gradient >25mmHg or aortic valve area <1.5cm²) and left ventricular ejection fraction >50%.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Combined outcome of death and cardiovascular-related hospitalization (including aortic valve replacement) | up to 10 years

SECONDARY OUTCOMES:
Combined outcome of death and cardiovascular-related hospitalization (without aortic valve replacement) | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Erwan Donal, MD, PhD, Study Chair — European Association of Cardiovascular Imaging
Locations (1):
- CHU LImoges, Limoges, France